CLINICAL TRIAL: NCT03690362
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of VNRX-5133 With VNRX-5022 in Subjects With Varying Degrees of Renal Impairment
Brief Title: VNRX-5133 With VNRX-5022 in Subjects With Varying Degrees of Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Venatorx Pharmaceuticals, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VNRX-5133-104; 272201300019C-12-0-3 (NIH); 17-0103 (Other: DMID)
Record Dates: First submitted 2018-03-21; First posted 2018-10-01 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — taniborbactam

STUDY DESIGN:
Intervention Model Description: The study will enroll approximately 32 subjects assigned to treatment groups based on renal function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 - Control (Experimental): Healthy control subjects will be matched by gender, weight, and age to subjects with renal impairment
  Interventions: Drug: VNRX-5133 and VNRX-5022
- Group 2 - Mild Renal Impairment (Experimental): Mild renal impairment
  Interventions: Drug: VNRX-5133 and VNRX-5022
- Group 3 - Moderate Renal Impairment (Experimental): Moderate Renal Impairment
  Interventions: Drug: VNRX-5133 and VNRX-5022
- Group 4 - Severe Renal Impairment (Experimental): Severe Renal Impairment
  Interventions: Drug: VNRX-5133 and VNRX-5022
- Group 5 - ESRD (Experimental): End Stage Renal Disease undergoing chronic intermittent hemodialysis
  Interventions: Drug: VNRX-5133 and VNRX-5022

INTERVENTIONS:
Drug: VNRX-5133 and VNRX-5022 — intravenous infusion

SUMMARY:
This is a multi-center, open-label, PK and safety study of VNRX-5133 and VNRX-5022 when co-administered in male and female subjects with varying levels of renal impairment and healthy normal controls.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18.5-40.0 kg/m2 with a minimum weight of 45 kg
* Able and willing to abstain from alcohol from 48 h before admission until the follow-up visit
* Suitable veins for cannulation/multiple venipunctures, as assessed by the Investigator at Screening
* Males who are not surgically sterilized and females of childbearing potential must agree to use highly effective methods of contraception during the study and for 90 days after study drug administration.
* Laboratory values meeting defined entry criteria

Subjects with normal renal function (Group 1) must also meet the following criteria:

* Match to one or more subjects with renal impairment by gender, age, and weight

Subjects with renal impairment (Groups 2-5) must also meet the following criteria:

* Stable, pre-existing renal impairment.

Exclusion Criteria:

* Employee of the study site, Contract Research Organization (CRO) or the IND Sponsor
* Female who is pregnant, lactating, or planning to attempt to become pregnant during the study or within 90 days after study drug administration
* Male with a female partner who is pregnant or lactating during the study, or planning to attempt to become pregnant during the study or within 90 days after study drug administration
* Use of any investigational drug or device within 30 days before study drug administration (90 days for an injectable biological agent)
* The subject has a congenital or acquired immunodeficiency syndrome
* Screening or Day -1, clinically significant abnormal ECG values
* Active malignancy; exceptions are permitted for carcinoma in situ of the prostate or the skin (basal cell or squamous cell) are permitted
* History of drug allergy of a severity that required urgent medical treatment, such as treatment with epinephrine in an Emergency Department
* Known immediate hypersensitivity reaction following administration of a cephalosporin, penicillin, or other β-lactam antibacterial drug
* History of donation of more than 450 mL of blood within 60 days before dosing in the site or planned donation before 30 days has elapsed since ingestion of study drug
* Plasma or platelet donation within 7 days of dosing and throughout the study
* Consumes more than 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of hard liquor) or has a significant history of alcohol abuse or drug/chemical abuse within the last 1 year
* Oral temperature >38.5˚C or acute illness on Day -1
* Previous participation in a study of VNRX-5133
* Excluded concomitant medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 72 hours
  To assess the pharmacokinetics of VNRX-5133 and VNRX-5022 in combination by assessment of Cmax
Area under the plasma concentration versus time curve (AUC) | 72 hours
  To assess the pharmacokinetics of VNRX-5133 and VNRX-5022 in combination by assessment of AUC
Safety and tolerability of VNRX-5133 and VNRX-5022 measured as number of subjects with adverse events. | 8 Days
  Number of Subjects with AEs (Assessed via patient report, physical exam, ECGs, vital signs, laboratory investigations, and use of concomitant medications for the treatment of AEs)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orlando Cliniical Research Associates, Orlando, Florida
  - New Orleans Center for Clinical Research, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dowell JA, Marbury TC, Smith WB, Henkel T. Safety and Pharmacokinetics of Taniborbactam (VNRX-5133) with Cefepime in Subjects with Various Degrees of Renal Impairment. Antimicrob Agents Chemother. 2022 Sep 20;66(9):e0025322. doi: 10.1128/aac.00253-22. Epub 2022 Aug 3. PMID 35920662